CLINICAL TRIAL: NCT01835652
Title: The Effects of Exercise in Parkinson's Disease.
Acronym: PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Parkinson's Research Centre (Other)
Responsible Party: Principal Investigator, A. Jon Stoessl, Director, Pacific Parkinson's Research Centre, Pacific Parkinson's Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H13-00276
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease 10
Keywords: Exercise; Parkinson's Disease; Positron Emission Tomography; fMRI
MeSH Terms: conditions — Parkinson Disease 10; Motor Activity; Parkinson Disease | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Exercise (Active Comparator): Aerobic Exercise Intervention (stationary cycling)
  Interventions: Other: Active Exercise
- Passive Exercise (Other): Passive Exercise (stretching and balance based exercise)
  Interventions: Other: Passive Exercise

INTERVENTIONS:
Other: Active Exercise
  Arms: Active Exercise
Other: Passive Exercise
  Arms: Passive Exercise

SUMMARY:
Parkinson's disease is caused by a reduction of dopamine causing motor deficits. The investigators are studying how exercise can help PD patients by increasing dopamine release in an area of the brain that coordinates movement, the striatum. The investigators will enroll PD patients into two groups; one group will complete a 12-week aerobic exercise program and the other will complete a 12-week control program including yoga and stretching only. The investigators will measure changes in dopamine release before and after either 12-week intervention. Subjects will complete motor and cognitive questionnaires in addition to functional magnetic resonance imaging and positron emission tomography neuroimaging.

DETAILED DESCRIPTION:
The purpose of this study is to determine the basis for symptomatic and disease modifying benefits of exercise in Parkinson's disease (PD).

Although the benefits of exercise in PD have been purported for several decades, only recently have there been controlled reports of symptomatic benefits in Parkinson's disease in terms of bradykinesia, postural balance and quality of life. There have been unsubstantiated suggestions that exercise may improve cognition and mood in PD.

The mechanisms underlying such benefits are poorly understood. Exercise may induce dopamine release, thereby contributing to improved motor function in the dorsal striatum, and to enhanced mood and reduced apathy in the ventral striatum.

We will test the hypotheses that exercise results in altered synaptic plasticity in the form of altered connectivity in response to aerobic exercise and reward-induced dopamine release. We will assess networks of functional connectivity using functional magnetic resonance imaging and measure dopamine release with positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD according to UK Brain Bank criteria (modified to permit inclusion of subjects with a family history)
2. Ages 40-70
3. Mild to moderate Parkinsonism (Hoehn & Yahr stages I-III)

Exclusion Criteria:

General exclusion criteria will include:

1. more than 120 minutes per week of activities >3 MET or a score exceeding 4 on the "Baseline Exercise Screening Tool" (Appendix, Fig. 1);
2. atypical Parkinson syndrome (progressive supranuclear palsy, multiple system atrophy, drug-induced etc.);
3. significant osteoporosis or arthritis;
4. other neurological disease (e.g. myopathy);
5. self-reports claustrophobia;
6. history of cancer within 5 years of study participation;
7. high dose of radiation from other procedures within the year;
8. taking rasagiline or selegiline for PD therapy;
9. diabetic;
10. not able to tolerate being off PD medication for up to 24 hours;
11. BMI of 35 or more; and
12. a female subject who is breast-feeding or pregnant.

Exclusion criteria for MRI scanning and magnetic stimulation from rTMS scanning includes:

1. artificial heart valve;
2. brain aneurysm clip;
3. electrical stimulator for nerves or bones;
4. ear or eye implant;
5. implanted drug infusion pump;
6. coil, catheter, or filter in any blood vessel;
7. orthopedic hardware (artificial joint, plate, screws);
8. other metallic prostheses;
9. shrapnel, bullets, or other metal fragments;
10. surgery or tattoos (including tattooed eyeliner) in the last six weeks;
11. have a cardiac pacemaker, wires or defibrillator;
12. have had an injury where a piece of metal lodged in your eye or orbit;
13. have a ferromagnetic aneurysm clip; and
14. have a history of seizures.

Subjects may be excluded following study enrollment if they meet any of the following exclusion criteria:

1. significant cognitive impairment (Montreal Cognitive Assessment score < 24) or depression (Beck Depression Inventory score > 18);
2. significant or unstable cardiovascular or respiratory disease - all subjects will undergo a screening exercise bicycle stress test; or
3. failure to comply with the exercise or yoga/stretching intervention program, including missing 5 sessions or missing three sessions in a row.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
PET | 3 months
  Dopamine release will be assessed using positron emission tomography (PET)

SECONDARY OUTCOMES:
fMRI | 3 months
  fMRI will be performed to record response to rewarding stimuli

OTHER OUTCOMES:
Clinical Measures | 3 months
  Motor function will be assessed using the MDS-Unified Parkinson's Disease Rating Scale, finger tapping and Purdue Pegboard. Cognitive function will be assessed using the Montreal Cognitive Assessment, Wisconsin Card-Sorting Task, Trail-Making B Test and a computerized reaction time test. Mood and apathy will be assessed using the Beck Depression Inventory and Starkstein Apathy Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jessamyn McKenzie, Study Director — Pacific Parkinson's Research Centre
Locations (1):
- Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886